CLINICAL TRIAL: NCT01148706
Title: Phase IV Study of the ActiSight Needle Guidance System Which Assist in Guiding a Rigid Interventional Instrument Percutaneously, to a Designated Point Within the Body by Means of CT Visualization
Brief Title: Effectiveness of ActiSight™ Needle Guidance System in Patients Undergoing CT-Guided Procedures
Acronym: ASNG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASNG-LFNA-103-IL
Record Dates: First submitted 2010-06-20; First posted 2010-06-22 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Lung Diseases; Liver Diseases
Keywords: thorax; abdomen
MeSH Terms: conditions — Lung Diseases; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ActiSight Needle Guidance System (Experimental)
  Interventions: Device: ActiSight Needle Guidance System

INTERVENTIONS:
Device: ActiSight Needle Guidance System — The ActiSight™ Needle Guidance System employs a miniature video camera mounted on the needle and a reference pad attached to the skin to register the needle into the CT image space, and thus, track the needle advance towards the target. CT scans are used as needed to verify the location of the needle.
  Other Names: ASNG=ActiSight Needle Guidance System

SUMMARY:
To assist in guiding a rigid interventional instrument percutaneously, to a designated point within the body by means of CT visualization.

DETAILED DESCRIPTION:
The ActiSight™ Needle Guidance System is an optical navigation system designed to assist physicians performing percutaneous interventions under CT guidance. The system allows the user to select an obstacle free path to a target lesion based on pre-procedure CT images, and then provides real-time information for guiding the interventional tool towards the target along the selected path.

The ActiSight™ Needle Guidance System employs a miniature video camera mounted on the needle and a reference pad attached to the skin to register the needle into the CT image space, and thus, track the needle advance towards the target. CT scans are used as needed to verify the location of the needle.

The primary objective of this study is to demonstrate the effectiveness of the ActiSight™ Needle Guidance System in assisting in CT-guided percutaneous procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment.
* Subjects meeting all medical conditions for percutaneous CT guided. procedures in the chest, abdomen or pelvic, with safe path to lesion.
* Written informed consent to participate in the study.
* Ability to comply with the requirements of the study procedures.

Exclusion Criteria:

* Having co-morbidities that would clinically preclude them from an image guided procedure as determined by the operating physician.
* Significant coagulopathy that cannot be adequately corrected.
* Patients who have a medical contraindication to sedation (Lidocaine allergy).
* Pregnancy or lactation.
* Participation in an investigational trial within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of CT scans performed during the procedure, from needle insertion to final needle position in the target lesion | 1 Hour- During the procedure

SECONDARY OUTCOMES:
Procedure time (needle dwell time in the body) | 1 hour -duration of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Natan Peled, Dr., Principal Investigator — Carmel MC
Locations (1):
- Carmel Medical Center, Haifa, Israel